CLINICAL TRIAL: NCT02829398
Title: Hemodynamic and Biochemical Determinants of Vasospasm and Delayed Ischemic Deficits in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Determinants of Vasospasm and Delayed Ischemic Deficits in Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07 304 02; Local Grant (Other Grant/Funding Number: 07 304 02)
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Ischemia
Keywords: cerebral ischemia
MeSH Terms: conditions — Ischemia; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with subarachnoid hemorrhage (Experimental): Patients with subarachnoid hemorrhage will have CerebroSpinal fluid and plasma sample.
  Interventions: Procedure: CerebroSpinal fluid and plasma samples
- Control subjects (Active Comparator): healthy controls from a previous study with a CerebroSpinal fluid and plasma sample
  Interventions: Procedure: CerebroSpinal fluid and plasma samples

INTERVENTIONS:
Procedure: CerebroSpinal fluid and plasma samples — CerebroSpinal fluid and plasma samples for biological markers

SUMMARY:
The risk of delayed cerebral ischemia (DCI) after subarachnoid hemorrhage (SAH) is associated with large cerebral artery vasospasm, but vasospasm is not a strong predictor for DCI. Assessment of cerebral autoregulation with transcranial Doppler (TCD) may improve the prediction of DCI. The aim of this prospective study was to assess the value of TCD-derived variables to be used alone or in combination for prediction of DCI

ELIGIBILITY:
Inclusion Criteria:

Group 1 : • Patients who presented a ruptured aneurysm by aneurysmal subarachnoid hemorrhage (SAH) older than 72 hours. Diagnosis of SAH was confirmed by computed tomography, magnetic resonance imaging (MRI) or lumbar puncture as recommended

* symptomatic aneurysm treated with endovascular,
* Absence of achieving a lumbar puncture,
* Patients affiliated to a social security scheme,
* Patients who have given their free and informed consent and signed the consent or consent of the family.

Group 2 :

healthy volunteers with cerebrospinal fluid sample

Exclusion Criteria:

* Patients with no readable acoustic temporal bone window
* Patients with previous disease that might impair cerebral autoregulation (e.g., carotid stenosis, history of stroke or head injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
delayed cerebral ischemia | inclusion
  DCI was confirmed by CT or MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: LARRUE Vincent, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calviere L, Nasr N, Arnaud C, Czosnyka M, Viguier A, Tissot B, Sol JC, Larrue V. Prediction of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage Using Cerebral Blood Flow Velocities and Cerebral Autoregulation Assessment. Neurocrit Care. 2015 Oct;23(2):253-8. doi: 10.1007/s12028-015-0125-x. PMID 25716738